CLINICAL TRIAL: NCT04440969
Title: Dementia - Early Detection and Intervention
Brief Title: Evaluation of Pilot Community-based Multi-domain Program Older Adults at Risk of Cognitive Impairment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Geriatric Education and Research Institute (Other Government)
Collaborators: Ministry of Health, Singapore (Other Government); Neeuro Pte Ltd (Unknown); ProAge Pte Ltd (Unknown); KKT Technology Pte Ltd (Holmusk) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: GERI1613; MOH/NIC/COG02/2017 (Other Grant/Funding Number: MOH)
Record Dates: First submitted 2020-06-16; First posted 2020-06-22 (Actual); Last update posted 2020-06-22 (Actual); Status verified 2020-06

CONDITIONS: Cognitive Decline; Cognitive Impairment, Mild
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Intervention administered is bi-weekly dual-task exercises, small group acitivites and computerised cognitive training for a total of 24 weeks. (Week 1 - 24)
  Interventions: Behavioral: Multi-domain intervention
- Wait-list control (Experimental): Intervention administered is bi-weekly dual-task exercises, small group acitivites and computerised cognitive training for a total of 24 weeks after Intervention Group has completed intervention. (Week 25 - 48)
  Interventions: Behavioral: Multi-domain intervention

INTERVENTIONS:
Behavioral: Multi-domain intervention — Participants will undergo dual-task physical exercises and small group activities comprising of quizzes, puzzles and simulate daily living activities that have been gamified (Mindfun and MindGym, ProAge,Singapore). They will also play games on a touch screen device (computerised cognitive training) that aims to improve cognition in the domains of attention, memory, spatial ability, decision making and cognitive flexibility (Memorie, Neeuro, Singapore) while wearing the Senzeband, which emits low frequency signals on the forehead picked up by four individual sensors, allowing participant to play certain games without touching the device but by attention and focus (https://www.neeuro.com/senzeband).
  Dietary guidance will be delivered via a dietary app (Glycoleap). Participants are expected to take photos of their meals daily and upload them onto the app. Certified dieticians will give advice and tips on their choice of food and how to make healthier choices through the app.

SUMMARY:
The multi-domain programme was adapted from a larger international multi-domain interventional study for the Singapore community of older adults at risk of cognitive impairment. This programme comprises nutritional, physical and cognitive components delivered by implementation partners in the community. A dementia risk screening tool developed from the Singapore Longitudinal Ageing Study (SLAS) data was used to screen potential participants. The nutritional component includes nutrition guidance via a nutritional app, while cognition component involves computerised training on a touch screen device and physical aspects involves dual-task exercises.

DETAILED DESCRIPTION:
Older people like to continue to think clearly, remember accurately, and make good decisions. The loss of the ability to live independently is one of the greatest fears adults express when considering old age. As physical fitness declines, the brain also ages. While cognition in areas related to wisdom and experience improve in older adults, others like memory, attention, and reaction time can decline and affect daily life. As life expectancy increases, maintaining cognition is critical to productive and healthy aging. Older adults want to continue to negotiate the environment, perform routine tasks (e.g. driving), learn new things, and live independently. Cognitive impairment creates significant challenges for individuals, their families and friends, and clinicians who provide their health care. Furthermore, available research indicates that cognitive impairment is not detected in substantial proportions of older people in primary care who have the condition. Early detection allows for earlier diagnosis and appropriate intervention, education, psycho-social support, and engagement in shared decision-making regarding life planning, financial matters, and health care. Based on this, there is a need for scalable, implementable intervention programmes which can be introduced in the community.

Previous studies have corroborated the efficacy of certain aspects of training which can promote delay in cognitive decline. Specifically, these encompass nutritional, cognitive and physical activity. Individually, these components have been extensively validated and proven effective in negating cognitive decline. However, little attempts have been made to evaluate the effectiveness and feasibility of combining these components into a multi-modal program. The only preceding study to have proven efficacy of multi-modal programs in improving cognition was carried out in the FINGER trial. However, to date, no similar studies have been carried out locally. Therefore, this study aims to address these questions; by using a mixed method approach; combining both qualitative and quantitative methods to assess the achievability of such a programme.

The programme aims to identify individuals at risk of cognitive decline and is offered to ensure intervention measures are adopted at early stages. The multi-domain program comprises a combination of nutritional guidance, group physical activity and cognitive training segments; all of which are individually regarded as proven interventions for cognitive impairment. The program will be coordinated between three commercial entities, Holmusk, Neeuro and ProAge and is funded by the National Innovation Challenge (NIC), MOH, Singapore. As part of the programme, the investigators will be utilizing a locally developed risk score created from the Singapore Longitudinal Aging study (SLAS), that can be widely administered and is applicable to the local population. Therefore, the study aims to use a mixed methods approach to evaluate:

1. The feasibility and sustainability of implementing the programme, which will be assessed based on several considerations such as reach, implementation and maintenance or areas of improvement.
2. The effectiveness of the programme on cognitive decline and improvement in fitness and nutrition.

ELIGIBILITY:
Inclusion Criteria:

* Above 55 years of age
* Interested & willing to participate in a lifestyle & cognition training programme
* Residing in Singapore over the next 1 year
* Have a risk score of more than 6-8, implying a 10-20% risk of developing cognitive decline over the next 5 years

Exclusion Criteria:

* Diagnosed with cognitive disorders such as mild cognitive impairment, dementia or Parkinson's Disease
* Wheelchair bound
* Total hearing or visual impairment
* Medical instructions prohibiting participation in the programme

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 199 (Actual)
Dates: Start 2018-06-20 (Actual); Primary Completion 2020-03-04 (Actual); Study Completion 2020-03-04 (Actual)

PRIMARY OUTCOMES:
Change from baseline in cognition at Week 12 and Week 48 | Baseline, Week 24 and Week 48
  Repeatable Battery for the Assessment of Neuropsychological Status (RBANS) is a cognitive test that consists of 12 subtests grouped into five domains - immediate and delayed memory, visuospatial/construction, language and attention. A higher score indicates better cognitive performance.

SECONDARY OUTCOMES:
Change from baseline in quality of life at Week 12 and Week 48 | Baseline, Week 24 and Week 48
  Quality of Life Questionnaire (EuroQol EQ-5D-5L) index measures participants' perception of their ability to 1) self-care, 2) carry out usual activities, and their levels of 3) mobility, 4) pain/discomfort, and 5) anxiety/depression. The EQ-5D index is derived by combining responses from these 5 categories. A higher index indicates higher quality of life. EQ-5D Visual Analogue Scale (VAS) is a 0 - 100 scale that measures participants' perception of their health status on the day this scale was used, with 100 signifying the best possible state of health.
Change from baseline in aerobic strength at Week 12 and Week 48 | Baseline, Week 24 and Week 48
  Two-minute step test is a test of aerobic endurance, where participants are required to take as many steps (marching on the spot) as possible in two minutes.
Change from baseline in leg strength at Week 12 and Week 48 | Baseline, Week 24 and Week 48
  Chair stand is a test of leg strength where participants are required to stand up from seated position as many times as possible in thirty seconds
Change from baseline in arm strength at Week 12 and Week 48 | Baseline, Week 24 and Week 48
  Handgrip strength is a test of hand and forearm muscular strength, where participants are required to squeeze a dynamometer as hard as possible. Units are measured in kilogrammes.

OTHER OUTCOMES:
Change from baseline in blood lipid levels at Week 12 and Week 48 | Baseline, Week 24 and Week 48
  Fasting blood sample collected via fingerprick to measure blood lipid levels on a rapid blood kit (Cholesh LDX, Abbott, IL, U.S)
Evaluation questionnaire | Week 24 and Week 48
  The questionnaire is to address some points of the REAIM framework, which stands for Reach, Effectiveness, Adoption, Implementation and Maintenance.
  Questions are either delivered on a 5-point Likert Scale for quantitative analysis (e.g.Did you find the exercises easy to follow? 1 - Extremely difficult, 2 - Quite difficult, 3 - Neutral, 4 - Quite easy, 5 - Extremely easy or as open ended questions for qualitative analysis (e.g. Are there barriers that will prevent you from taking up the programme?) Questionnaires are delivered to participants, centre managers and implementation partners.

CONTACTS AND LOCATIONS:
Overall Officials: Shiou Liang Wee, PhD, Principal Investigator — Geriatric Education and Research Institute
Locations (1):
- Geriatric Education And Research Institute, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No
Due to confidentiality issues, individual participant data will not be made public but de-identified data can be obtained upon request.

REFERENCES:
- [Background] Lustig C, Shah P, Seidler R, Reuter-Lorenz PA. Aging, training, and the brain: a review and future directions. Neuropsychol Rev. 2009 Dec;19(4):504-22. doi: 10.1007/s11065-009-9119-9. Epub 2009 Oct 30. PMID 19876740
- [Background] Morley JE, Morris JC, Berg-Weger M, Borson S, Carpenter BD, Del Campo N, Dubois B, Fargo K, Fitten LJ, Flaherty JH, Ganguli M, Grossberg GT, Malmstrom TK, Petersen RD, Rodriguez C, Saykin AJ, Scheltens P, Tangalos EG, Verghese J, Wilcock G, Winblad B, Woo J, Vellas B. Brain health: the importance of recognizing cognitive impairment: an IAGG consensus conference. J Am Med Dir Assoc. 2015 Sep 1;16(9):731-9. doi: 10.1016/j.jamda.2015.06.017. PMID 26315321
- [Background] Ahlskog JE, Geda YE, Graff-Radford NR, Petersen RC. Physical exercise as a preventive or disease-modifying treatment of dementia and brain aging. Mayo Clin Proc. 2011 Sep;86(9):876-84. doi: 10.4065/mcp.2011.0252. PMID 21878600
- [Background] Kivipelto M, Solomon A, Ahtiluoto S, Ngandu T, Lehtisalo J, Antikainen R, Backman L, Hanninen T, Jula A, Laatikainen T, Lindstrom J, Mangialasche F, Nissinen A, Paajanen T, Pajala S, Peltonen M, Rauramaa R, Stigsdotter-Neely A, Strandberg T, Tuomilehto J, Soininen H. The Finnish Geriatric Intervention Study to Prevent Cognitive Impairment and Disability (FINGER): study design and progress. Alzheimers Dement. 2013 Nov;9(6):657-65. doi: 10.1016/j.jalz.2012.09.012. Epub 2013 Jan 17. PMID 23332672
- [Background] Ngandu T, Lehtisalo J, Solomon A, Levalahti E, Ahtiluoto S, Antikainen R, Backman L, Hanninen T, Jula A, Laatikainen T, Lindstrom J, Mangialasche F, Paajanen T, Pajala S, Peltonen M, Rauramaa R, Stigsdotter-Neely A, Strandberg T, Tuomilehto J, Soininen H, Kivipelto M. A 2 year multidomain intervention of diet, exercise, cognitive training, and vascular risk monitoring versus control to prevent cognitive decline in at-risk elderly people (FINGER): a randomised controlled trial. Lancet. 2015 Jun 6;385(9984):2255-63. doi: 10.1016/S0140-6736(15)60461-5. Epub 2015 Mar 12. PMID 25771249
- [Background] Smith PJ, Blumenthal JA. Diet and neurocognition: review of evidence and methodological considerations. Curr Aging Sci. 2010 Feb;3(1):57-66. doi: 10.2174/1874609811003010057. PMID 20298171
- [Background] Rawtaer I, Feng L, Yuen VH, Li J, Chong MS, Lim WS, Lee TS, Qiu C, Feng L, Kua EH, Ng TP. A Risk Score for the Prediction of Neurocognitive Disorders among Community-Dwelling Chinese Older Adults. Dement Geriatr Cogn Disord. 2016;41(5-6):348-58. doi: 10.1159/000447448. Epub 2016 Jul 20. PMID 27433801
- [Derived] Ng PEM, Nicholas SO, Wee SL, Yau TY, Chan A, Chng I, Yap LKP, Ng TP. Implementation and effectiveness of a multi-domain program for older adults at risk of cognitive impairment at neighborhood senior centres. Sci Rep. 2021 Feb 15;11(1):3787. doi: 10.1038/s41598-021-83408-5. PMID 33589714